CLINICAL TRIAL: NCT05057091
Title: Immediate Effects of Two Spinal Manipulative Techniques on Clinical Outcomes and Muscle Mechanical Properties in Chronic Low Back Pain: An Assessor Blinded, Randomized Controlled Trial
Brief Title: Immediate Effects of Two Spinal Manipulative Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, pHd., Clinical Physiotherapist, Principal invetsigator, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10354421-2021/03-14
Record Dates: First submitted 2021-09-06; First posted 2021-09-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-back Pain
Keywords: Acute Manipulation; Chronic manipulation; Low back pain; muscles mechanical treshold; physiotherapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This research is planned as a double blind randomized controlled trials
Masking Description: A power analysis was conducted to determine the number of cases to be included in the study. In order for the study to be performed at 80% strength and with a 5% margin of error, at least 23 people from each group should be included in the study to find a difference of 30 N/m after application, in the case where the lumbal extensor November hardness is 320 N/m and the standard deviation is 74 N/m
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Maitland's Posterior-Anterior Central Vertebral Manipulation (Experimental): The posterior-anterior unilateral vertebral manipulation.
  Interventions: Other: Group 1 - Maitland's Posterior-Anterior Central Vertebral Manipulation; Other: Group 2- Side-Lying Lumbar Spinal Manipulation
- Group 2- Side-Lying Lumbar Spinal Manipulation (Experimental): A high-speed, low-amplitude thrust force was applied in opposite directions: anteriorly to the pelvis and posteriorly to the shoulder
  Interventions: Other: Group 1 - Maitland's Posterior-Anterior Central Vertebral Manipulation; Other: Group 2- Side-Lying Lumbar Spinal Manipulation

INTERVENTIONS:
Other: Group 1 - Maitland's Posterior-Anterior Central Vertebral Manipulation — For the posterior-anterior unilateral vertebral manipulation, the therapist positioned both thumbs on top of each other on the spinous process of the vertebra and applied an average of 4 kg of discrete pressure
Other: Group 2- Side-Lying Lumbar Spinal Manipulation — The therapist stood in front of the patient, who was instructed to lie on their side with the painful side facing upward.the therapist utilized their arm and body to apply the manipulation. A high-speed, low-amplitude thrust force was applied in opposite directions: anteriorly to the pelvis and posteriorly to the shoulder.

SUMMARY:
The aim of this study is to investigate the instant effects of direct vertabral manipulation and indirect vertebral manipulation techniques on muscles mechanical properties, pressure-pain threshold and joint range of motion in individuals with chronic low back pain. Another purpose of this study was to compare the effects of both treatment methods on the parameters studied.

DETAILED DESCRIPTION:
Resolving chronic low back pain is a costly obstacle. There is a wide spectrum of treatment for chronic low back pain, such as exercise training, pain training and spinal manipulation.It is the recommended spinal manipulation in the short and long term in chronic low back pain. Clinical Spinal manipulation is one of the most preferred methods of reducing pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 ages
* Individuals with non-specific chronic low back pain who have continued pain for at least 3 months
* According to VAS, individuals with pain of at least 3 severity

Exclusion Criteria:

* Pregnancy situation or suspicion
* Spinal Stenosis
* Vertebral fracture
* Cancer
* Osteoporosis
* Individuals with BMI over 30 kg/m2
* Those with neurological disease that leads to November loss of muscle strength or spasticity-rigidity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Mechanical properties measurements | through study completion, an average of 1 hour
  A MyotonPro was used to measure the mechanical properties of selected muscles. the measurements of the medial gastrocnemius and biceps femoris muscles were performed while individuals were in prone position the knees at full extension, and the ankle at neural position. The measurements of medial gastrocnemius were performed on plumped portion of the muscle at a point 70% of the lower leg length in line with the popliteal crease to the lateral malleolus. For biceps femoris muscle, measurements were performed at the middle points between tuberosity of the ischium and the head of the fibula.the mechanical properties of lumbar extensor muscle were performed while the individuals were prone position the hip and knee at full extension. For lumbar extensor muscle, the measurements were performed at the point 3 cm from the midpoint of the L3/L4 intervertebral space. The average of three consecutive measurements was recorded.

SECONDARY OUTCOMES:
Oswestry low back pain scale | Through study completion, an average of 1 hour
  it measures a total of 10 different aspects, severity of pain, personal care, lifting, walking, sitting, standing, sleeping, degree of pain change, social life, travel to assess the effect of low back pain on daily life activities in the patient.
Roland morris disability scale | Through study completion, an average of 1 hour
  This questionnaire is a 24-point questionnaire designed to assess the degree of functional limitation in patients with low back pain. In the survey, the answers vary from yes to no yes: 1 point, no: 0 points, and high scores indicate severe obstacle status
Visual analog scale | Through study completion, an average of 1 hour
  VAS was used to measure the severity of the patient's pain. It is usually 10 cm long, horizontal or vertical; it is a line that begins with "no pain" and ends with "unbearable pain". This line can only be a straight line, or divided into equal December, or in pain definition, the definition placed on the line can be found in words. The patient indicates the severity of his pain with a sign where he sees fit on this line. "Cm" was measured and recorded between the point marked with the onset of decontamination. "0 'means no pain,' 5 'means moderate pain,' 10" means the most severe pain encountered in life.
Fear Avoidance Beliefs Questionnare | Through study completion, an average of 1 hour
  Fear avoidance beliefs questionnare has 16 questions and two sub-scales, physical activity and work. The physical activity section consists of 5 questions, and the work section consists of 11 questions. The survey was a Likert-type scale of 7. In the answers given to the survey, the expression I disagree with at all is given 0 points and the expression I fully agree with is given 6 points.

OTHER OUTCOMES:
Modify shober test | The measurements were performed before and immediately after the applications.
  Lumbal region flexion flexibility was measured by modified Schober Test.
Sit and reach tets | The measurements were performed before and immediately after the applications.
  Lumbar region extansors flexibilty test was measured by sit and reach test

CONTACTS AND LOCATIONS:
Overall Officials: Emine KURT, Assc. Prof., Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)